CLINICAL TRIAL: NCT03622788
Title: Anti-Viral Central Memory CD8 Veto Cells in Haploidentical Hematopoietic Stem Cell Transplantation
Brief Title: Cytokine-Treated Veto Cells in Treating Patients With Hematologic Malignancies Following Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0221; NCI-2018-01557 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0221 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-08-03; First posted 2018-08-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Aplastic Anemia; Bone Marrow Failure; Chronic Lymphocytic Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Follicular Lymphoma; Hodgkin Lymphoma; Mantle Cell Lymphoma; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Non-Hodgkin Lymphoma; Plasma Cell Myeloma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Aplastic; Bone Marrow Failure Disorders; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Follicular; Hodgkin Disease; Lymphoma, Mantle-Cell; Myelodysplastic Syndromes; Myeloproliferative Disorders; Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — Antilymphocyte Serum; Cyclophosphamide; fludarabine; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Treatment (chemotherapy, PBSCT, cytokine-treated veto cells) (Experimental): CONDITIONING REGIMEN: Patients receive ATG IV over 4 hours on days -9 to -7, and fludarabine IV over 1 hour on days -6 to -3, then undergo TBI on day -1.
  TRANSPLANT: Patients undergo PBSCT IV over 30-60 minutes on day 0.
  GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 3 hours on days +3 and +4 and cytokine-treated veto cells IV over 30-60 minutes on day +7.
  Interventions: Biological: Anti-Thymocyte Globulin; Drug: Cyclophosphamide; Biological: Cytokine-treated Veto Cells; Drug: Fludarabine; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Total-Body Irradiation

INTERVENTIONS:
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATS
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Cytokine-treated Veto Cells — Given IV
  Other Names: Activated Veto Cells; Activated Veto T-cells; Veto CD8-positive T-cells; Veto Cell; Veto Cells; Veto-enhanced CTL; Veto-enhanced Cytotoxic T-cell
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSCT
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; PERIPHERAL BLOOD STEM CELL TRANSPLANT; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: SCT_TBI; TBI; Total Body Irradiation; Whole Body Irradiation; Whole-Body Irradiation

SUMMARY:
This phase I/II trial studies how well cytokine-treated veto cells work in treating patients with hematologic malignancies following stem cell transplant. Giving chemotherapy and total-body irradiation before a stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the patient, they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Cytokine-treated veto cells may help the transplanted donor cells to develop and grow in recipients without causing graft-versus-host-disease (GVHD - when transplanted donor tissue attacks the tissues of the recipient's body).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the optimal dose of anti-viral veto cells, defined as the dose which achieves engraftment without severe graft-vs-host disease (GVHD) at 42 days after non-myeloablative megadose T cell depleted haploidentical hematopoietic cell transplantation (HCT).

SECONDARY OBJECTIVES:

I. Toxicity. II. Response rate. III. Time to progression. IV. Infections. V. Immune reconstitution. VI. Overall survival up to 1 year.

OUTLINE: This is a dose-escalation study of cytokine-treated veto cells.

CONDITIONING REGIMEN: Patients receive anti-thymocyte globulin (ATG) intravenously (IV) over 4 hours on days -9 to -7 and fludarabine IV over 1 hour on days -6 to -3, then undergo total body irradiation (TBI) on day -1.

TRANSPLANT: Patients undergo peripheral blood stem cell transplantation (PBSCT) IV over 30-60 minutes on day 0.

GVHD PROPHYLAXIS: Patients receive cyclophosphamide IV over 3 hours on days +3 and +4 and cytokine-treated veto cells IV over 30-60 minutes on day +7.

After completion of stem cell transplant, patients are followed up once a week for 4 weeks, once a month for 3 months, and then periodically for one year.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age 12-75 years. The first 3 subjects will be 18 years of age to gain experience and observe safety. After 3 adult subjects have successfully engrafted and if the safety profile is tolerable, adolescents age 12 may be enrolled on to the trial
* Patients with a diagnosis either follicular lymphoma (FL), mantle cell lymphoma (MCL), chronic lymphocytic leukemia (CLL), multiple myeloma (MM), Hodgkin's lymphoma (HL), non-Hodgkin's lymphoma (NHL), chronic myeloid leukemia (CML), myelodysplastic syndrome, myeloproliferative syndromes (MPD), acute myeloid leukemia (AML) or acute lymphoid leukemia (ALL).
* Patients with aplastic anemia and severe immune deficiency or nonmalignant bone marrow failure states. Patients with severe thalassemia requiring regular blood transfusions or sickle cell disease with severe clinical features (these include any clinically significant sickle genotype, for example, hemoglobin SS (Hb SS), hemoglobin SC (Hb SC), hemoglobin S beta thalassemia (Hb Sbeta), or Hemoglobin S-OArab genotype] with at least one of the following manifestations:

  * Clinically significant neurologic event (stroke) or neurological deficit lasting > 24 hours;
  * History of two or more episodes of acute chest syndrome (ACS) in the 2-year period preceding enrollment or referral despite adequate supportive care measures (i.e. asthma therapy);
  * An average of three or more pain crises per year in the 2-year period preceding enrollment or referral (required intravenous pain management in the outpatient or inpatient hospital setting);
  * Administration of regular red blood cell (RBC) transfusion therapy, defined as 8 or more transfusion events per year (in the 12 months before enrollment) to prevent vaso-occlusive clinical complications (i.e. pain, stroke, or acute chest syndrome);
  * An echocardiographic finding of tricuspid valve regurgitant jet (TRJ) velocity >= 2.7 m/sec.
  * Ongoing high impact1 chronic pain on a majority of days per month for >= 6 months as defined as ONE or more of the following: Chronic pain without contributory sickle cell disease (SCD) complications2, OR mixed pain type in which chronic pain is occurring at site(s) (arms, back, chest, or abdominal pain) unrelated to any sites associated with contributory SCD complications2 (e.g. leg ulcers and/or avascular necrosis)
* Patients with hematological malignancies must have had persistent or progressive disease despite initial chemotherapy and must have achieved stable disease or a partial or complete response to their most recent chemotherapy. Patients with low bulk or indolent relapse are eligible without additional treatment. Patients with high-risk acute myeloid leukemia by European LeukemiaNet (ELN) criteria in first remission are eligible.
* Availability of a medically acceptable haploidentical related donor, age 12-70 years.
* Karnofsky performance status >= 70%.
* Left ventricular ejection fraction of at least 40%.
* Pulmonary function test (PFT) demonstrating an adjusted diffusion capacity of least 50% predicted value for hemoglobin concentration.
* Serum creatinine =< 1.5 mg/dl.
* Serum glutamic-pyruvic transaminase (SGPT) =< 200 IU/ml.
* Bilirubin < 1.5 mg/dl (unless Gilbert's syndrome).
* Negative pregnancy test in a woman with childbearing potential.

Patient Exclusion Criteria:

* Human immune deficiency virus (HIV) seropositive.
* Uncontrolled infection or serious medical or psychiatric condition that would limit tolerance to the protocol treatment.
* Active central nervous system (CNS) malignancy.
* Availability of medically eligible, human leukocyte antigen (HLA)-matched related stem cell donor.

Donor Inclusion Criteria

* Medically acceptable haploidentical donor age 12-70 years.
* Hemoglobin > 12.0 g/dL [female] or > 13.0 g/dL [male] or > 11.0 g/dL for females of childbearing potential with documented iron deficiency anemia
* Platelet count 150, 0000/ul
* WBC 3.0 - 11.0 K/ul
* No anomalies on CBC and differential indicating a hematopoietic disorder
* Negative pregnancy test for women of childbearing potential; Not lactating
* Systolic blood pressure < 170 mmHg and Diastolic blood pressure < 95 mmHg
* Performance status KPS > 70%
* CXR negative for active infection or malignancy
* EKG not suggestive of uncontrolled cardiac disease
* No known allergy to cytokines if cytokines are to be used.
* No active or uncontrolled autoimmune disorders
* Completion and signature of donor questionnaire (within 30 days)
* Donor infectious disease panel and health assessment performed by attending physician

Donor Exclusion Criteria

* Individuals with cognitive impairments and/or any serious unstable pre-existing condition or psychiatric disorder that can interfere with safety or without obtaining informed consent or compliance with study procedures.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Optimal dose of donor-derived cytokine-treated veto cells | Within 42 days of cytokine-treated veto cell infusion
  For the purpose of dose-finding, toxicity is defined as steroid resistant grade 3 or 4 graft-versus-host-disease (GVHD), or death from any cause, within 42 days of veto cell infusion.
Efficacy of veto cells | At day 42 post cytokine-treated veto cell infusion
  Efficacy is defined as the patient being alive and engrafted at day 42 post veto cell infusion.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 1 year
  Unadjusted distributions of time-to-event outcomes will be estimated using the method of Kaplan and Meier and their relationship to prognostic covariates and veto cell dose level will be evaluated by Bayesian piecewise exponential survival regression.
Response rate | Up to 1 year
  Unadjusted distributions of time-to-event outcomes will be estimated using the method of Kaplan and Meier and their relationship to prognostic covariates and veto cell dose level will be evaluated by Bayesian piecewise exponential survival regression.
Time to progression | Up to 1 year
  Unadjusted distributions of time-to-event outcomes will be estimated using the method of Kaplan and Meier and their relationship to prognostic covariates and veto cell dose level will be evaluated by Bayesian piecewise exponential survival regression.
Infections | Up to 1 year
  Unadjusted distributions of time-to-event outcomes will be estimated using the method of Kaplan and Meier and their relationship to prognostic covariates and veto cell dose level will be evaluated by Bayesian piecewise exponential survival regression.
Immune reconstitution | Up to 1 year
  Unadjusted distributions of time-to-event outcomes will be estimated using the method of Kaplan and Meier and their relationship to prognostic covariates and veto cell dose level will be evaluated by Bayesian piecewise exponential survival regression.
Overall survival | Up to 1 year
  Unadjusted distributions of time-to-event outcomes will be estimated using the method of Kaplan and Meier and their relationship to prognostic covariates and veto cell dose level will be evaluated by Bayesian piecewise exponential survival regression.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Champlin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org